CLINICAL TRIAL: NCT06509971
Title: A Study of QL1706 (an Anti-PD-1/CTLA-4 Combined Antibody) Combined With Albumin-bound Paclitaxel and Bevacizumab in the Treatment of Platinum-resistant Recurrent Ovarian Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: West China Second University Hospital (Other)
Responsible Party: Principal Investigator, Rutie Yin, Head of chemoradiotherapy department, West China Second University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WCSUH20240707
Record Dates: First submitted 2024-07-07; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Platinum-resistant Recurrent Ovarian Cancer
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): QL1706: 5 mg/kg Q3W, IV , up to 34 courses.
  Albumin-binding paclitaxel: 260 mg/m2 Q3W, IV, 6 courses.
  Bevacizumab: 15 mg/kg Q3W, IV, up to 22 courses.
  Interventions: Drug: QL1706

INTERVENTIONS:
Drug: QL1706 — The Order of Drug Administration was: QL1706→ bevacizumab → albumin-binding paclitaxel, and each drug was administered at least 30 minutes apart.
  QL1706: 5 mg/kg Q3W. The infusion time was 30 minutes + 5 minutes. No dose adjustment was allowed for QL1706 during treatment, but delayed administration was allowed, with a delay of no more than 4 weeks from the previous dose.
  Albumin-binding paclitaxel: 260 mg/m 2 Q3W, IV, for 30 min + 5 min. During treatment, albumin-binding paclitaxel allows for dose adjustments.
  Bevacizumab: 15 mg/kg Q3 W, iv. The first infusion should last 90 minutes. If the first infusion was well tolerated, the second infusion could be shortened to 60 minutes. If the patient is also well-tolerated for a 60-minute infusion, then all subsequent infusions can be completed in 30 minutes, no dose adjustment is allowed for bevacizumab.
  Other Names: bevacizumab; albumin-binding paclitaxel

SUMMARY:
* Major objectives To evaluate the efficacy of QL1706 combined with albumin-binding paclitaxel and bevacizumab in the treatment of platinum-resistant recurrent ovarian cancer.
* Secondary Purpose To evaluate the safety of QL1706 in combination with albumin-binding paclitaxel and bevacizumab in the treatment of platinum-resistant recurrent ovarian cancer.

Exploratory analysis of the association between the efficacy of the combination regimen and biomarkers.

DETAILED DESCRIPTION:
The efficacy of chemotherapy combined with anti-angiogenic agents in the treatment of platinum-resistant recurrent ovarian cancer has been demonstrated in clinical studies, and QL1706 acts as a bi-functional combination antibody that blocks both PD-1 and CTLA-4, in other cancer trials that have been conducted, it is expected that better efficacy and adverse event rates comparable to those of anti-PD-1 mabs and anti-CTLA-4 mabs will be achieved with combination chemotherapy and anti-angiogenic drugs, it may be possible to obtain better anti-tumor effects in platinum-resistant recurrent ovarian cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary signing of a written ICF.
2. Age ≥18 years, ≤75 years, female.
3. The Eastern Cooperative Oncology Group (ECOG) physical fitness score was 0 or 1.
4. Expected survival ≥3 months.
5. Histologically or cytologically confirmed epithelial ovarian cancer, fallopian tube cancer, or primary peritoneal cancer.
6. Patients with platinum-resistant recurrent ovarian cancer (including fallopian tube and peritoneal cancer) were defined as progression within 6 months after platinum-based chemotherapy.
7. At least one measurable lesion according to RECIST v1.1, and this lesion is amenable to repeated accurate measurements according to RECIST v1.1. Lesions that have received radiation therapy can be considered as target lesions if they are clearly progressive and measurable on the basis of imaging.
8. Determination of good organ function through the following requirements:

   A) hematology (no blood component and cell growth factor support therapy was used for 7 days before study initiation) :

   I. ANC ≥1.5 × 109 L (1.500 MM3) in absolute neutrophil; II. Platelet count ≥100 × 109/L (100,000/MM3) ; III. Hemoglobin ≥90 g/L.

   B) kidneys:

   I. Creatinine clearance * (CrCl) calculated value ≥50 mL/min

   * CrCl (Cockcroft-gault formula) will be calculated using Cockcroft-Gault formula CrCL (mL/min) = [(140-age) × weight (kg) × f ]/(SCR (mg/dL) × 72) F = 0.85; SCR = serum creatinine. II. Urine protein < 2 + or 24 h (h) urine protein quantification < 1.0 g.

   C) liver:

   I. Serum total bilirubin (TBil)≤1.5 × ULN II. AST and ALT ≤2.5 × ULN III. Alb (Alb)≥28GL

   D) coagulation function:

   I. International standard ratio (INR) and activated partial thromboplastin time (APTT)≤1.5 × ULN.

   E) cardiac function:

   I. Left ventricular ejection fraction (LVEF)≥50% .
9. A fertile female subject must have a urine or serum pregnancy test within 3 days before the first dose (if the urine pregnancy test result can not be confirmed as negative, a serum pregnancy test is required, whichever is the serum pregnancy result) , and the results were negative. If a fertile female subject has sex with an unsterilized male partner, the subject must use an acceptable method of contraception from the beginning of the screening process, consent must also be given to the method of contraception used prior to its continued use for 120 days after the last administration of the study drug; discontinuation of contraception after this time point should be discussed with the investigator.
10. Subjects were willing and able to comply with schedule visits, treatment protocols, laboratory tests, and other requirements of the study.

Exclusion Criteria:

1. Ovarian cancer of non-epithelial origin, fallopian tube cancer, primary peritoneal cancer (such as germ cell tumors) , and low-malignant potential ovarian tumors (such as borderline tumors) .
2. Previous (within 5 years) or concurrent with other malignancies, the local tumors that have been cured (such as basal cell skin cancer, squamous cell skin cancer, superficial bladder cancer, cervical carcinoma in situ, breast carcinoma in situ, etc.) and breast cancer that has not recurred for more than 3 years after radical operation are excluded.
3. Local recurrence is suitable for patients undergoing surgery.
4. Previous radiation therapy of the abdomen and pelvis.
5. Had received immunotherapy in the past, these include immune-checkpoint inhibitors (such as PD-1 CTLA-4 Bispecific monoclonal antibody, which allow previous use of PD-1 or PD-L1 mabs) , immune-checkpoint agonists (such as ICOS, CD40, CD137, GITR, OX40 antibodies, etc.) , and immune-cell therapies for any of the mechanisms of tumor immunity.
6. Patients who were known to be allergic to any component of any investigational drug, had a history of severe hypersensitivity to other monoclonal antibody, and were known to have permanently discontinued the relevant therapeutic drug could not be enrolled.
7. Participated in the treatment of an experimental drug or used an experimental device within 4 weeks before the first study administration.
8. One week before the first dose (or 5 drug half-lives, whichever is longer) , a potent or intermediate CYP3A4 inhibitor, a P-gp or a BCRP inhibitor were received.
9. Last systemic anti-tumor therapy, including chemotherapy, bevacizumab or its bioanalogues, was given within 3 weeks before the first dose, and anti-tumor hormone therapy was given within 2 weeks before the first dose Non-target lesions were treated with palliative local therapy within 2 weeks before the first dose Received Hapten therapy (such as interleukin, interferon, and thymosin, not including Il-11 for thrombocytopenia) within 2 weeks before the first dose; Within 1 week before the first administration, she had received Chinese herbal medicine or Chinese patent medicine with anti-tumor indication.
10. Use of systemic glucocorticoid or other immunosuppressive drug within one week prior to initial administration, systemic glucocorticoid (i.e. not more than 10mg daily prednisone or equivalent dose of other glucocorticoid) that do not include nasal spray, inhalation or other route local glucocorticoid or physiological doses, allow for symptoms of dyspnea due to diseases such as chronic obstructive pulmonary disease, and temporary use of glucocorticoid for allergy prevention.
11. The live vaccine was administered within 30 days of the first dose, or was planned for the duration of the study.
12. Has an active autoimmune disease that requires systemic treatment in the past two years (such as use of disease-modifying drugs, corticosteroid, immunosuppressive therapy) , replacement therapy (such as thyroxine, insulin, or physiologic corticosteroid for adrenal or pituitary insufficiency) is not considered a systemic treatment.
13. Active or previous history of a well-defined inflammatory bowel disease such as Crohn's disease, ulcerative colitis or chronic diarrhea.
14. History of immunodeficiency, HIV antibody positive, current long-term use of systemic corticosteroid or other immunosuppressive agents.
15. Subjects with known active tuberculosis (TB) and suspected active TB should be excluded by clinical examination.
16. Known active syphilis infection.
17. Known history of organ transplants and Hematopoietic stem cell transplants.
18. Previous history of non-infectious pneumoniainterstitial lung disease requiring systemic glucocorticoid therapy or current presence of non-infectious pneumonia.
19. Severe infection occurred within 4 weeks before the first dose, including but not limited to complications, sepsis, or severe pneumonia requiring hospitalization; Active infection (excluding antiviral therapy for hepatitis B or C) that has received systemic anti-infective therapy within 2 weeks before the first dose.
20. Untreated subjects with active hepatitis B (HBsAg positive and HBV-DNA > 1000 copies/ml (200 IU/ml or above the lower limit of detection, whichever is higher) were required to receive anti-hbv therapy during study treatment for those with hepatitis B; and active hepatitis C subjects (HCV antibody positive and HCV-rna levels above the lower limit of detection) .
21. Those who had a major surgical procedure or major trauma within 30 days before the first dose, or who had a major surgical plan within 30 days after the first dose (at the investigator's discretion) ; Minor local procedures (excluding central venous catheterization via peripheral venipuncture and intravenous port implantation) were performed within 3 days before the first dose.
22. Known presence of central nervous system metastases, meningeal metastases, spinal cord metastases or compression.
23. Subjects with clinical symptoms or repeated drainage of pleural effusion, pericardial effusion, or ascites.
24. There are currently uncontrolled co-morbidities, these include, but are not limited to, symptomatic heart failure (grade 2 or higher according to the New York Heart Association functional class) , unstable angina, acute myocardial ischemia, poorly controlled arrhythmias, decompensated cirrhosis, nephrotic syndrome, uncontrolled metabolic disorders, severe active peptic ulcer disease, or gastritis, psychiatric/social conditions that may limit subjects' ability to comply with research requirements or affect their ability to provide written informed consent.
25. Uncontrolled hypertension, systolic blood pressure > 140 mmhg or diastolic blood pressure > 90 mmhg after optimal medical treatment, history of Hypertensive crisis or hypertensive encephalopathy.
26. Previous history of myocarditis, cardiomyopathy, and malignant arrhythmia. Unstable angina, myocardial infarction, heart failure or vascular disease (such as a ruptured aortic aneurysm) that requires hospitalization within 12 months of the first dose, or other cardiac lesions (such as poorly controlled arrhythmias, myocardial ischemia) that may affect the safety evaluation of the study drug.
27. Esophageal Gastric varices, severe ulcers, unhealed wounds, gastrointestinal perforation, abdominal fistula, gastrointestinal obstruction, intra-abdominal abscess, acute gastrointestinal bleeding, extensive bowel resection (partial or extensive colectomy with chronic diarrhea) , Crohn's disease, ulcerative colitis or chronic diarrhea.
28. Any arterial thromboembolic event, NCI CTCAE version 5.0 Grade 3 or greater, venous thromboembolism, transient cerebral ischemia, or cerebrovascular accident occurred within 6 months before the first dose.
29. Acute exacerbation of chronic obstructive pulmonary disease within 1 month of first dose.
30. Patients with any sign of bleeding constitution, regardless of severity; patients with any bleeding or bleeding event ≥ CTCAE grade 3 within 4 weeks before the first dose.
31. Current imaging or clinical manifestations of gastrointestinal obstruction, including incomplete obstruction.
32. Severe bleeding tendency or Coagulopathy, or receiving thrombolytic therapy. Aspirin (> 325mg daily) or dipyrimidine, ticlopidine, clopidogrel, and Cilostazol are currently used or have been used recently (within 10 days before the first dose of study treatment) , and anticoagulants that require monitoring of INR (such as Warfarin) .
33. Imaging showed that the tumor had surrounded or invaded important blood vessels, or that it was highly likely to invade important blood vessels and cause fatal massive bleeding during the follow-up study, compression of the superior vena cava, inferior vena cava or invasion of the heart.
34. Toxicities from previous antitumour therapy did not resolve, defined as toxicities that did not return to grade 0 or 1 of NCI CTCAE version 5.0, or levels specified in the inclusion/exclusion criteria; Except for alopecia and sequelae of neurotoxicity related to previous platinum therapy. For subjects who develop irreversible toxicity and are not expected to worsen after administration of the study drug (EG, hearing loss) , it may be included in the study after consultation with the medical examiner.
35. Local or systemic disease caused by a non-malignant tumor, or disease or symptoms secondary to the tumor, and can lead to higher medical risk and/or uncertainty in the evaluation of survival; Such as leukemoid reaction cancer (white blood cell count > 20 × 10 ^ 9 L) , cachexia (known as weight loss of more than 10% 3 months before screening) , etc. .
36. Known history of mental illness, substance abuse, alcohol or drug abuse.
37. Women who are pregnant or nursing. The presence of any disease, treatment, or laboratory abnormality in the past or present may confuse the results of the study, affect the participant's participation in the study, or may not be in the best interest of the participant.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 6 months
  Defined as the proportion of subjects achieving optimal total efficacy (Bor) as confirmed Cr or PR (according to RECIST v1.1) . The best overall response was defined as the best response recorded (in order of CR, PR, SD, PD, or non-evaluable) from the beginning of treatment until disease progression, or in cases where PD was not achieved before the initiation of subsequent antitumour therapy or before study discontinuation (whichever occurred first) , the best efficacy was recorded (from the start of treatment until the last evaluable tumour imaging assessment) .

IPD SHARING:
Plan to Share IPD: Undecided